CLINICAL TRIAL: NCT03386097
Title: Studies of the Importance of Interstitial Fluid in the Development of Cardiovascular Disease, an Expanded Study.
Brief Title: Interstitial Fluid in the Development of Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Mats Rudling, Professor, MD, Karolinska University Hospital
Other Study IDs: DiabetesIC2
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Type2 Diabetes; Atherosclerosis
Keywords: Cholesterol; Interstitial fluid
MeSH Terms: conditions — Atherosclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Interstitial fluid, skin biopsies and blood (serum, plasma and whole blood)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 diabetes patients
  Interventions: Other: Collection of interstitial fluid, skin biopsies and blood
- Healthy controls
  Interventions: Other: Collection of interstitial fluid, skin biopsies and blood

INTERVENTIONS:
Other: Collection of interstitial fluid, skin biopsies and blood — Collection of interstitial fluid, skin biopsies and blood

SUMMARY:
At a given level of serum cholesterol, patients with T2D have an increased risk of developing atherosclerosis compared with nondiabetic subjects.

In a previous study we showed that the interstitial fluid-to-serum gradient of LDL and VLDL cholesterol is reduced in T2D patients compared with healthy controls. This was not found for HDL cholesterol. However, the cholesterol transporting function of HDL particles from interstitial fluid from patients with T2D were lower than in healthy controls. We hypothesize that that the apo B-containing particles in T2D patients are more susceptible to be retained or consumed in the extravascular space.

We are to study if skin biopsies from T2D patients contain more cholesterol than biopsies from healthy controls. We hypothesize that samples from T2D patients are richer in cholesterol, which could explain why VLDL and LDL cholesterol are lower in relation to their plasma levels in T2D.

ELIGIBILITY:
Inclusion criteria:

* Over 18 years.
* For the T2D study group: Diagnosed with type 2 diabetes.

Exclusion criteria:

For subjects with type 2 diabetes:

* Systemic inflammatory disease that requires active treatment
* Thyroid disease that requires active treatment
* Skin disease that requires active treatment and causes significant changes in the area of the skin that is to be investigated
* Treatment with oral glucocorticoids
* Levels of SR, TSH, T4 or Hemoglobin in the blood pronouncedly outside the reference range
* Pregnancy

For healthy controls:

* Registered disease in the health declaration that requires continuous systemic treatment. Exception to the above: well controlled hypertension in which case the subject should not have treatment with more than one antihypertensive drug, the drug must not be an alpha-blocker or beta-blocker or thiazide diuretic
* Skin disease that requires active treatment and causes significant changes in the area of the skin that is to be investigated
* Blood pressure pronouncedly above 140/90
* Blood test results pronouncedly outside the reference range
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls and type 2 diabetes patients over 18 years old, matched for age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Interstitial fluid-to-serum ratio for LDL cholesterol | 2 hours
Cholesterol level in skin biopsies | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mats Rudling, Principal Investigator — Karolinska Institutet
Locations (4):
- Sweden (4):
  - Ekerö Vårdcentral, Ekerö, Ekerö Kommun
  - Patient research centre, Clinic of endocrinology, Karolinska University Hospital, Huddinge, Stockholm County
  - Stiftelsen Stockholms Sjukhems Husläkarmottagning, Stockholm
  - GIH (gymnastik och idrottshögskolan), Stockholm

IPD SHARING:
Plan to Share IPD: No